CLINICAL TRIAL: NCT03227796
Title: A Randomised, Double-blind, Placebo-controlled, Single Ascending Dose, Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of LEVI-04 in Healthy Volunteers and Patients With Pain Attributed to Osteoarthritis of the Knee
Brief Title: Safety, Tolerability & Pharmacokinetics of LEVI-04 in Healthy Volunteers and Patients With Osteoarthritis Knee Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Levicept (Industry)
Collaborators: Hammersmith Medicines Research (Other); MAC Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: LEVI-04_17_01
Record Dates: First submitted 2017-05-31; First posted 2017-07-24 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Healthy Volunteers; Osteoarthritis
Keywords: osteoarthritis; knee; healthy; volunteer; LEVI-04
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: First-in-human, phase 1, placebo-controlled, double-blind, single ascending dose study in heathy volunteers and osteoarthritis patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (16):
- Cohort 1 Healthy Volunteers Active (Experimental): LEVI-04 0.003 mg/kg single intravenous dose Healthy Volunteers
  Interventions: Drug: LEVI-04
- Cohort 2 Healthy Volunteers Active (Experimental): LEVI-04 Dose Level 2 (planned 0.01 mg/kg) single intravenous dose Healthy Volunteers
  Interventions: Drug: LEVI-04
- Cohort 3 Healthy Volunteers Active (Experimental): LEVI-04 Dose Level 3 (planned 0.03 mg/kg) single intravenous dose Healthy Volunteers
  Interventions: Drug: LEVI-04
- Cohort 4 Osteoarthritis Patients Active (Experimental): LEVI-04 Dose Level 3 (planned 0.03 mg/kg) single intravenous dose Osteoarthritis Patients
  Interventions: Drug: LEVI-04
- Cohort 5 Osteoarthritis Patients Active (Experimental): LEVI-04 Dose Level 4 (planned 0.1 mg/kg) single intravenous dose Osteoarthritis Patients
  Interventions: Drug: LEVI-04
- Cohort 6 Osteoarthritis Patients Active (Experimental): LEVI-04 Dose Level 5 (planned 0.3 mg/kg) single intravenous dose Osteoarthritis Patients
  Interventions: Drug: LEVI-04
- Cohort 7 Osteoarthritis Patients Active (Experimental): LEVI-04 Dose Level 6 (planned 1.0 mg/kg) single intravenous dose Osteoarthritis Patients
  Interventions: Drug: LEVI-04
- Cohort 8 Healthy Volunteers Active (Experimental): LEVI-04 Dose Level 7 (planned 3.0 mg/kg) single intravenous dose Healthy Volunteers
  Interventions: Drug: LEVI-04
- Cohort 1 Healthy Volunteers Placebo (Placebo Comparator): Placebo to match LEVI-04 single intravenous dose Healthy Volunteers
  Interventions: Drug: Placebo
- Cohort 2 Healthy Volunteers Placebo (Placebo Comparator): Placebo to match LEVI-04 single intravenous dose Healthy Volunteers
  Interventions: Drug: Placebo
- Cohort 3 Healthy Volunteers Placebo (Placebo Comparator): Placebo to match LEVI-04 single intravenous dose Healthy Volunteers
  Interventions: Drug: Placebo
- Cohort 4 Osteoarthritis Patients Placebo (Placebo Comparator): Placebo to match LEVI-04 single intravenous dose Osteoarthritis Patients
  Interventions: Drug: Placebo
- Cohort 5 Osteoarthritis Patients Placebo (Placebo Comparator): Placebo to match LEVI-04 single intravenous dose Osteoarthritis Patients
  Interventions: Drug: Placebo
- Cohort 6 Osteoarthritis Patients Placebo (Placebo Comparator): Placebo to match LEVI-04 single intravenous dose Osteoarthritis Patients
  Interventions: Drug: Placebo
- Cohort 7 Osteoarthritis Patients Placebo (Placebo Comparator): Placebo to match LEVI-04 single intravenous dose Osteoarthritis Patients
  Interventions: Drug: Placebo
- Cohort 8 Healthy Volunteers Placebo (Placebo Comparator): Placebo to match LEVI-04 single intravenous dose Healthy Volunteers
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LEVI-04 — LEVI-04 intravenous infusion
  Arms: Cohort 1 Healthy Volunteers Active; Cohort 2 Healthy Volunteers Active; Cohort 3 Healthy Volunteers Active; Cohort 4 Osteoarthritis Patients Active; Cohort 5 Osteoarthritis Patients Active; Cohort 6 Osteoarthritis Patients Active; Cohort 7 Osteoarthritis Patients Active; Cohort 8 Healthy Volunteers Active
Drug: Placebo — Placebo intravenous infusion
  Arms: Cohort 1 Healthy Volunteers Placebo; Cohort 2 Healthy Volunteers Placebo; Cohort 3 Healthy Volunteers Placebo; Cohort 4 Osteoarthritis Patients Placebo; Cohort 5 Osteoarthritis Patients Placebo; Cohort 6 Osteoarthritis Patients Placebo; Cohort 7 Osteoarthritis Patients Placebo; Cohort 8 Healthy Volunteers Placebo

SUMMARY:
This is a first-in-human, phase 1, single centre, placebo-controlled, double-blind, single ascending dose study of LEVI-04 in heathy volunteers and osteoarthritis patients (with pain attributed to osteoarthritis of the knee)

DETAILED DESCRIPTION:
There will be 8 cohorts of 7 subjects each. Cohorts 1-3 and 8 will be composed of healthy volunteers. Cohorts 4-7 will be composed of osteoarthritis patients. Cohort 4 will be a bridging cohort; osteoarthritis patients in Cohort 4 will receive the same dose as the healthy volunteers in Cohort 3, if deemed safe.

Each subject will be assigned to receive a single dose of LEVI-04 or matching placebo. Each dose will be administered as an intravenous infusion over 30 minutes. Planned doses will start at 0.003 mg/kg in Cohort 1, and may be increased to 3.0 mg/kg in Cohort 8. The planned doses may be changed, depending on the safety, tolerability and pharmacokinetic results after previous doses. The dose selected for each cohort will be determined by the Safety Review Team, following review of all available pharmacokinetic and safety data. For each escalating dose, there will be at least 2 weeks between the start of each cohort (at least 14 days between Day 0 for the last subject in the previous cohort and Day 0 for the first subject in the subsequent cohort), to allow for review of safety, tolerability and pharmacokinetic data. In each cohort, 5 subjects will receive LEVI-04 and 2 subjects will receive matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.0-<32.0 kg/m2 (healthy volunteers) and 18.0-<40.0 kg/m2 (osteoarthritis patients)
* Willing and able to give written fully informed consent
* Men with female partners of childbearing potential must agree to follow the requirements for effective contraception throughout the study and for 112 days post-dose
* Women of non childbearing potential
* Healthy volunteers (aged 18 to 65 years) willing to give written consent to have data entered into the Over-volunteering Prevention System
* Osteoarthritis patients (aged 30-80 years) with diagnosis of mild to moderate osteoarthritis of the knee, with X-ray confirmation as diagnosed by a trained radiology reviewer
* Osteoarthritis patients willing to discontinue all pain medication, except rescue medication (paracetamol), from the run-in visit until the end of the study
* Osteoarthritis patients with a Numerical Rating Scale-11 pain score of between 5 and <9, inclusive, in the index knee at screening. If taking regular pain medication, should show an increase of at least 1 point following washout of analgesia. The average pain score of between 5 and <9, inclusive, based on four of the seven daily readings during the seven day initial pain assessment period

Exclusion Criteria:

* Women of childbearing potential, or who are pregnant or lactating
* Clinically relevant abnormal history, physical findings, electrocardiograph, or laboratory values at screening that could interfere with the objectives of the trial or the safety of the subject
* Presence of acute or chronic illness or history of chronic illness (other than osteoarthritis, controlled diabetes, asthma or hypertension for osteoarthritis patients), sufficient to invalidate participation in the trial or make it unnecessarily hazardous
* Impaired endocrine, thyroid, hepatic, respiratory (other than asthma that has been controlled by the use of acceptable medication for at least 3 months prior to screening) or renal function; or history of any psychotic mental illness or clinically significant psychiatric disorder
* History of carpal tunnel syndrome with signs or symptoms within one year before screening or a Boston Carpal Tunnel Questionnaire score >3
* Moderate or severe carpal tunnel syndrome based on the 4th finger neurological test or Total Neuropathy Score nurse
* History of cancer within 5 years before screening, except for appropriately treated cutaneous basal cell or squamous cell cancers; cervical cancer; and low grade stable prostate cancer
* History, diagnosis, or signs of neurological disease including but not limited to: stroke; peripheral or autonomic neuropathy; diabetic neuropathy; multiple sclerosis; epilepsy or seizure disorder with history of seizure within last 2 years; myopathy; Alzheimer's disease or other types of dementia; head trauma within last 2 years; and episodic lower limb radiculopathy, nerve compression, or sciatica (provided diagnosed as due to nerve root compression and not as a manifestation of systemic neuropathy or radiculopathy)
* Survey of Autonomic Symptoms score of at least 3
* Uncontrolled type 1 diabetes or type 2 diabetes with HbA1c <7.5% (type 1 diabetics and type 2 diabetics that have been controlled by acceptable medication for at least three months prior to screening are permitted if HbA1c < 7.5%).
* History or signs and symptoms of coronary heart disease or stroke
* QTcF interval <330 msec or ≥430 msec for males, and ≥450 msec for females at the screening examination, unless judged not clinically significant by an investigator
* Presence of Chronic Obstructive Pulmonary Disease
* Moderate / severe depression indicated by a score of ≥10 out of 24 in the Personal Health Questionnaire Depression Scale
* History or presence of severe adverse reaction to any drug or a history of sensitivity to mannitol or histidine
* Use of prescription medicine (other than the permitted medicines) during 28 days before the dose of trial medication (14 days for pain medication for osteoarthritis patients)
* Use of an over-the-counter medicine, except paracetamol, during the 7 days before the first dose of trial medication
* Dosed in another clinical trial of a new chemical entity or prescription medicine within last 3 months
* Previous use of any Tropomyosin-receptor kinase (TrkA) inhibitor, Nerve Growth Factor-targeted therapy (eg tanezumab), or experimental biological treatment in last 6 months. More than 6 doses of anti- nerve growth factor (NGF) antibody during participation in a trial is not permitted.
* History / presence of drug / alcohol abuse in year before screening, or intake of >28 units of alcohol weekly or currently smoking >10 cigarettes daily
* Evidence of drug abuse
* Uncontrolled hypertension (supine) at screening outside 90-140 mm Hg systolic, 40-90 mm Hg diastolic; heart rate in supine position at screening outside 40-100 beats/min. (Diagnosed hypertension that has been controlled within the above limits using acceptable medication for at least 3 months prior to screening is permitted.)
* Possibility that will not cooperate with requirements of the trial
* Positive test for hepatitis B, hepatitis C or Human Immunodeficiency Virus
* Loss of more than 400mL blood during last 3 months, eg as a blood donor
* Objection by General Practitioner to trial entry
* Poor venous access

Also for osteoarthritis patients:

* History of inflammatory arthritis, including rheumatoid arthritis, seronegative spondyloarthropathy (eg ankylosing spondylitis, psoriatic arthritis, inflammatory bowel disease related arthropathy), gout, pseudogout in index knee (as diagnosed by appropriate crystals on aspiration or C-reactive protein elevation during attacks (subjects with gout or pseudogout in a joint other than the index knee must have disease that is controlled by medication, with a serum uric acid within the target range; should their index knee flare up during the study, gout must be excluded), metabolic joint disease, endocrinopathy, lupus erythematosus, joint infection, connective tissue disease, septic arthritis
* Radiographic evidence of:

  * excessive malalignment of the knee
  * severe chondrocalcinosis or other arthropathies (eg rheumatoid arthritis)
  * systemic metabolic bone disease (eg pseudogout, Paget's disease, metastatic calcifications)
  * large cystic lesions, primary or metastatic tumour lesions
  * acute or healing stress or traumatic fracture (subjects with established united/ malunited intra or extra-articular fractures of the knee from historic injuries [>12 months prior to screening] who have developed features of post-traumatic osteoarthritis can be included in the trial, provided that clinically and radiologically there is no excessive malalignment of the knee)
  * Rapidly Progressive Osteoarthritis, or any condition which would indicate an increased risk for developing it
  * atrophic or hypotrophic osteoarthritis
  * subchondral insufficiency fractures
  * spontaneous osteonecrosis of the knee
  * osteonecrosis
  * pathologic fracture
* History of osteonecrosis / osteoporotic fracture (including minimally traumatic or atraumatic fracture)
* History of significant trauma (including sports injury) or surgery to a knee, hip or shoulder within last year
* Planned surgery to a knee, hip or shoulder during the study
* Fibromyalgia, regional pain caused by lumbar / cervical compression with radiculopathy, or other moderate/severe pain that may confound assessment of knee pain
* Intra-articular injection of corticosteroid in the index knee within 3 months, or to any other joint within 1 month of the initial pain assessment
* Intra-articular injection of any hyaluronan product in the index knee within 6 months before the initial pain assessment
* Any other medical or psychiatric condition, or laboratory abnormality, that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the investigator would make the subject inappropriate for entry into this study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events [Safety and tolerability] | Change from Baseline at Day 56 post-dose for healthy volunteers and change from Baseline at Day 105 post-dose for osteoarthritis patients
  adverse events; laboratory tests; electrocardiograms and injection site reaction assessments
Change from Baseline in neurological assessments [Safety and tolerability] - SAS | Change from Baseline at Day 56 post-dose for healthy volunteers and change from Baseline at Day 105 post-dose for osteoarthritis patients
  Neurological assessment (Survey of Autonomic Symptoms (SAS) Questionnaire)
Change from Baseline in neurological assessments [Safety and tolerability] - BCTQ | Change from Baseline at Day 56 post-dose for healthy volunteers and change from Baseline at Day 105 post-dose for osteoarthritis patients
  Neurological assessment (Boston Carpal Tunnel Questionnaire (BCTQ)
Change from Baseline in neurological assessments [Safety and tolerability] - 4th finger test | Change from Baseline at Day 56 post-dose for healthy volunteers and change from Baseline at Day 105 post-dose for osteoarthritis patients
  Neurological assessment (the carpal tunnel syndrome (CTS) 4th finger neurological test or Total Neuropathy Score nurse)

SECONDARY OUTCOMES:
Pharmacokinetics of single ascending intravenous doses of LEVI-04 in healthy volunteers and osteoarthritis patients - maximum concentration | Up to Day 56 post-dose for healthy volunteers and up to Day 105 post-dose for osteoarthritis patients
  Maximum serum concentration
Pharmacokinetics of single ascending intravenous doses of LEVI-04 in healthy volunteers and osteoarthritis patients - time to maximum concentration | Up to Day 56 post-dose for healthy volunteers and up to Day 105 post-dose for osteoarthritis patients
  Time to reach maximum serum concentration
Pharmacokinetics of single ascending intravenous doses of LEVI-04 in healthy volunteers and osteoarthritis patients - Area Under the Curve | Up to Day 56 post-dose for healthy volunteers and up to Day 105 post-dose for osteoarthritis patients
  Area under the serum concentration-time curve from time zero to time of last measurable concentration
Pharmacokinetics of single ascending intravenous doses of LEVI-04 in healthy volunteers and osteoarthritis patients - half-life | Up to Day 56 post-dose for healthy volunteers and up to Day 105 post-dose for osteoarthritis patients
  Terminal elimination half-life
Pharmacokinetics of single ascending intravenous doses of LEVI-04 in healthy volunteers and osteoarthritis patients - clearance | Up to Day 56 post-dose for healthy volunteers and up to Day 105 post-dose for osteoarthritis patients
  Apparent total body clearance after intravenous administration
Pharmacokinetics of single ascending intravenous doses of LEVI-04 in healthy volunteers and osteoarthritis patients - elimination rate | Up to Day 56 post-dose for healthy volunteers and up to Day 105 post-dose for osteoarthritis patients
  Terminal elimination rate constant
Pharmacokinetics of single ascending intravenous doses of LEVI-04 in healthy volunteers and osteoarthritis patients - volume of distribution | Up to Day 56 post-dose for healthy volunteers and up to Day 105 post-dose for osteoarthritis patients
  Apparent volume of distribution during the terminal elimination phase
To assess the formation of anti-drug antibodies (ADA) to LEVI-04 in healthy volunteers and osteoarthritis patients | Up to Day 56 post-dose for healthy volunteers and up to Day 105 post-dose for osteoarthritis patients
  Presence / concentration of any anti-drug antibodies to LEVI-04

OTHER OUTCOMES:
Pharmacodynamics of LEVI-04 in osteoarthritis patients - pain relief (rescue medication) | Up to Day 105 for osteoarthritis patients
  Use of rescue medication, by treatment and time point
Pharmacodynamics of LEVI-04 in osteoarthritis patients - pain relief (NRS-11) | Up to Day 105 for osteoarthritis patients
  Assessment of pain using the Numerical Rating Scale-11 (NRS-11) questionnaire by treatment and time point
Pharmacodynamics of LEVI-04 in osteoarthritis patients - pain relief (WOMAC) | Up to Day 105 for osteoarthritis patients
  Assessment of pain using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire by treatment and time point
Exploratory analyses of pharmacological biomarkers relevant to the actions of LEVI-04 in healthy volunteers and osteoarthritis patients (NGF) | Up to Day 56 post-dose for healthy volunteers and up to Day 105 for osteoarthritis patients
  Measurement of total, free and LEVI-04 bound Nerve Growth Factor (NGF)
Exploratory analyses of pharmacological biomarkers relevant to the actions of LEVI-04 in healthy volunteers and osteoarthritis patients (NT-3) | Up to Day 56 post-dose for healthy volunteers and up to Day 105 for osteoarthritis patients
  Measurement of Neurotropin-3 (NT-3)

CONTACTS AND LOCATIONS:
Overall Officials: Denisa Wilkes, MUDr, Principal Investigator — Hammersmith Medicines Research
Locations (2):
- United Kingdom (2):
  - MAC Clinical Research - Early Phase Unit, Manchester, Greater Manchester
  - Hammersmith Medicines Research, London

IPD SHARING:
Plan to Share IPD: No